CLINICAL TRIAL: NCT02879825
Title: Myocardial Characterization of Arrhythmogenic Mitral Valve Prolapse
Brief Title: Myocardial Characterization of Arrhythmogenic Mitral Valve Prolapse (STAMP: STretch and Myocardial Characterization in Arrhythmogenic Mitral Valve Prolapse)
Acronym: STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Olivier HUTTIN, Medical Doctor, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00954-47
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Mitral Valve Prolapse
Keywords: Ventricular Premature Complexes
MeSH Terms: conditions — Mitral Valve Prolapse; Ventricular Premature Complexes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Mitral valve prolapse without mitral regurgitation
  Interventions: Device: Cardiac MRI
- Group B (Experimental): Mitral valve prolapse with trivial mitral regurgitation
  Interventions: Device: Cardiac MRI
- Group C (Experimental): Mitral valve prolapse with moderate or mild mitral regurgitation and asymptomatic
  Interventions: Device: Cardiac MRI
- Group D (Experimental): Mitral valve prolapse with severe mitral regurgitation or symptomatic
  Interventions: Device: Cardiac MRI

INTERVENTIONS:
Device: Cardiac MRI — Group-A patients, with mitral valve prolapse but no mitral regurgitation, will undergo specifically for research purposes a cardiac MRI, 24-hour external loop recording and exercise ECG on top of regular echocardiography evaluation.
  Realization of these examinations will be performed according to recommendations for patients with mitral regurgitation (groups B, C and D)
  Other Names: 24-hour external loop recording; Exercise ECG

SUMMARY:
Mitral valve prolapse (MVP) is a frequent affection of the mitral valve or its sub-valvular apparatus with a prevalence of 2-3% in the general population. This valvular disease is generally considered as benign, but may at term evolve toward mitral valve regurgitation of various severity and/or arrhythmia.

Mitral valve prolapse is routinely diagnosed using transthoracic echocardiography and only patients with significant mitral regurgitation will undergo subsequent examination (24-hour external loop recording, exercise ECG, cardiac MRI) and a close follow-up.

External loop recording and exercise ECG have an interest in the identification of patients presenting with arrhythmic complications, such as premature ventricular contractions, and in the global evaluation of hemodynamic consequences of the mitral regurgitation.

More recently, detection of myocardial fibrosis among patients with MVP and severe ventricular arrhythmia has been identified. Fibrosis could evolve independently of the valvular regurgitation's severity and could be a substrate (myocardial scar) leading to ventricular arrhythmia. However, no study has specifically characterized myocardial lesions among patients with MVP and none, or not significant, mitral regurgitation. Using cardiac magnetic resonance imaging (MRI), gold standard technique in myocardial imaging and characterization, and echocardiography, particularly speckle-tracking imaging, identification of static (fibrosis) and/or dynamic (ventricular systolic deformation patterns using speckle-tracking strain) myocardial lesions.

Identification of patients with impaired deformation patterns, fibrosis or with premature ventricular contractions may isolate a sub-group of patients with a higher risk of severe ventricular arrhythmia for whom a closer follow-up could be justified.

ELIGIBILITY:
Inclusion Criteria:

* Mitral valve prolapse diagnosed in echocardiography
* Signed written consent
* Affiliation to social security
* No contraindication to MRI or exercise ECG
* Age above 18

Exclusion Criteria:

* Mitral valve prolapse with severe regurgitation and instable hemodynamic state requiring urgent surgery
* Prior MRI with contrast within the last month
* Prior diagnosis of primary cardiomyopathy potentially responsible for myocardial fibrosis
* Contraindication to exercise ECG: severe handicap, poor physical capacity
* Contraindication to MRI: implantable device, claustrophobia, metal debris
* Renal insufficiency with creatinine clearance <30 ml/min or prior serious side effect related to infusion of a magnetic contrast agent
* Pregnant or breast-feeding women
* Minors <18 years old
* Mental illness or incapacity with incapacity to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Evidence of ventricular arrythmia (premature ventricular contraction or tachycardia) | Within 15 days
  Occurrence of any ventricular arrythmia on external loop recording or exercise ECG
Evidence of myocardial fibrosis on cardiac MRI | Within 15 days
  Visualisation of any late gadolinium enhancement

SECONDARY OUTCOMES:
Estimation of mitral regurgitation severity on echocardiography | At inclusion
Description and evaluation of ventricular myocardial deformation patterns | Within 15 days
  Comparison of deformation patterns using speckle-tracking echocardiography and strain in cardiac MRI
Comparative evaluation of mitral regurgitation using echocardiography and cardiac MRI | Within 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HUTTIN, MD, MSc, Principal Investigator — Department of Cardiology, Nancy University Hospital
Locations (1):
- Nancy University Hospital, Department of Cardiology, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Basso C, Perazzolo Marra M, Rizzo S, De Lazzari M, Giorgi B, Cipriani A, Frigo AC, Rigato I, Migliore F, Pilichou K, Bertaglia E, Cacciavillani L, Bauce B, Corrado D, Thiene G, Iliceto S. Arrhythmic Mitral Valve Prolapse and Sudden Cardiac Death. Circulation. 2015 Aug 18;132(7):556-66. doi: 10.1161/CIRCULATIONAHA.115.016291. Epub 2015 Jul 9. PMID 26160859
- [Background] Huttin O, Pierre S, Venner C, Voilliot D, Sellal JM, Aliot E, Sadoul N, Juilliere Y, Selton-Suty C. Interactions between mitral valve and left ventricle analysed by 2D speckle tracking in patients with mitral valve prolapse: one more piece to the puzzle. Eur Heart J Cardiovasc Imaging. 2017 Mar 1;18(3):323-331. doi: 10.1093/ehjci/jew075. PMID 27099279
- [Derived] Huttin O, Girerd N, Jobbe-Duval A, Constant Dit Beaufils AL, Senage T, Filippetti L, Cueff C, Duarte K, Fraix A, Piriou N, Mandry D, Pace N, Le Scouarnec S, Capoulade R, Echivard M, Sellal JM, Marrec M, Beaumont M, Hossu G, Trochu JN, Sadoul N, Marie PY, Guenancia C, Schott JJ, Roussel JC, Serfaty JM, Selton-Suty C, Le Tourneau T. Machine Learning-Based Phenogrouping in MVP Identifies Profiles Associated With Myocardial Fibrosis and Cardiovascular Events. JACC Cardiovasc Imaging. 2023 Oct;16(10):1271-1284. doi: 10.1016/j.jcmg.2023.03.009. Epub 2023 May 17. PMID 37204382